CLINICAL TRIAL: NCT01758510
Title: An Open-label, Phase 1 Trial for Safety Study of HLA-haplo Matched Allogenic Bone Marrow Derived Stem Cell("HYNR-CS-Allo Inj") Treatment in Amyotrophic Lateral Sclerosis(ALS)
Brief Title: Safety Study of HLA-haplo Matched Allogenic Bone Marrow Derived Stem Cell Treatment in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Corestemchemon, Inc. (Industry)
Responsible Party: Principal Investigator, Seung Hyun Kim, Professor/Dept. Neurology, College of Medicine, Hanyang University Seoul Hospital, Hanyang University Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYNR-CS-Allo-01
Record Dates: First submitted 2012-12-10; First posted 2013-01-01 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Disease; Neurodegenerative Disease; Central Nervous System Disease
Keywords: Amyotrophic Lateral Sclerosis; ALS; Neurodegenerative disease; Motor Neuron Disease; Central Nervous System Disease; Neuromuscular Disease; Bone marrow derived stem cell; stem cell therapy; intrathecal injection
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases; Neurodegenerative Diseases; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HYNR-CS-Allo (Experimental): HYNR-CS-Allo inj. 2 times by intrathecal administration with 28 days interval.
  Interventions: Genetic: HYNR-CS-Allo

INTERVENTIONS:
Genetic: HYNR-CS-Allo — The patients enrolled in the trial will be successively allocated into three cohorts for HYNR-CS-Allo inj., 0.25 X 10^6 cells/kg, 0.5 X 10^6 cells/kg, 1 X 10^6 cells/kg, according to the 3+3, up and down protocol design. The first treatment cohort will be 0.5 X 10^6 cells/kg dose cohort.

SUMMARY:
The purpose of this study is to evaluate the safety of HLA-haplo matched Allogenic Bone Marrow Derived stem cells("HYNR-CS-Allo inj"), through intrathecal delivery for the treatment in patients with amyotrophic lateral sclerosis(ALS).

This study is an open label, dose up and down study using the 3+3 design to assess the safety of HLA-haplo matched Allogenic Bone Marrow Derived stem cells("HYNR-CS-Allo inj")

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a progressive neurodegenerative disease characterized by motor neuron loss. Despite of many trials for disease-modifying, no treatment has so far changed natural course of disease.

The investigators had performed the pre-clinical and clinical studies using autologous bone marrow-derived stem cells in ALS. In the investigators' results of clinical trial, intrathecal injection of autologous bone marrow-derived stem cells is safe and could slow down disease progression and might be used as a disease modifying strategy in patients with ALS.

In the new field, like cell therapy, it is an important issue whether a bone marrow derived mesenchymal stem cells can be used as an allograft. Many investigators had showed that the immunoprivileged and immunosuppressive properties of mesenchymal stem cells result from the absence of major histocompatibility class II antigens and the secretion of T helper type 2 cytokines.

One potential advantage of allogenic bone marrow derived cells could be avoiding the need for procedural delay before treatment. And it is also hypothesized that the function of autologous bone marrow derived cells could be impaired in patients with co-morbidities or advanced age.

This study is to evaluate safety of HYNR-CS-Allo inj(HLA-haplo matched Allogenic bone marrow-derived stem cells) in patients with ALS.

The patients enrolled in the trial will be successively allocated into three cohorts for HYNR-CS-Allo inj., 0.25 X 10^6 cells/kg, 0.5 X 10^6 cells/kg, 1 X 10^6 cells/kg, according to the 3+3, up and down protocol design. The first treatment cohort will be 0.5 X 106 cells/kg dose cohort. Only a maximum of six patients will be given a particular dosage.

The scheduled assessments and visits will be carried out over three periods: run-in period, treatment period, and follow-up period.

The run-in period includes the screening visit where a written informed consent is obtained and the screening period where patients are assessed for eligibility. It will be completed within 30 days prior to enrollment. The patients meeting inclusion criteria will start the treatment period.

During the treatment period, subjects will be administered HYNR-CS-Allo inj. 2 times by intrathecal administration with 28 days interval.

The Follow-up period starts once subjects complete the treatment period and will continue until the final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 25 and 80 years old
* Patients who have both signs of lower motor neuron(LMN) and upper motor neuron(UMN) degeneration by clinical, electrophysiological or neuropathologic examination
* Patients diagnosed as 'Probable' or 'Definite' ALS according to the World Federation of Neurology El Escorial criteria
* Patients whose duration of disease is within 5 years from the first diagnosis
* Patients with ALSFRS-R score within 21 to 46 at screening
* Patients who can visit to a hospital by walk personally or by protector's help
* Patients who provide the written consent by oneself or his/her legal representative
* Patients who has HLA-haplo matched Bone marrow donor

Exclusion Criteria:

* Patients who doesn't appropriate to the diagnostic criteria of ALS
* Patients who are diagnosed as primary lateral sclerosis(PLS) or progressive muscular atrophy(PMA)
* Patients suspected of adverse effect after stem cell injection(patients suspected of malignant tumor, risk group of psychogenic shock, patients with serious hypertension)
* Patients with ALSFRS-R score below 21 at screening
* Patients performed ventilator or tracheostomy at screening
* Patients performed gastrostomy at screening
* Patients unable to assess the efficacy of this clinical trial due to unattainable Pulmonary Functional Test(PFT) or patients with suspected 40% or less of Forced vital capacity(FVC) at screening
* Patients with finding of myocardial infarction or angina pectoris according to ECG, patients who have been performed Stenting or Bypass operation at screening
* Patients who have taken any other drug for clinical trial within the past 3 months at screening entry
* Patients with epilepsy
* Patients with severe renal dysfunction(serum creatinine≥2.0mg/dl)
* Patients with severe liver dysfunction(ALT, AST, bilirubin≥upper limit of normal X 2)
* Pregnant woman, lactating woman, female patients who has a pregnancy planning or who doesn't agree with adoption of contraception methods proper medically, male patients who doesn't agree with adoption of contraception methods proper to his partner during participating this study
* Patients with hemorrhagic tendency at screening
* Patients with virus infection at screening
* Patients with a known history of hypersensitivity/allergy to penicillin and streptomycin
* Patients with previous stem cell therapy
* Patients diagnosed with cancer
* Patients who have taken any drug that can effect to bone marrow function
* Patients with any other neurological disease except ALS
* Patients with psychotic diseases

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events(SAE) | 6 months
  The Incidence of any treatment related serious adverse events(SAE)

SECONDARY OUTCOMES:
ALS-Functional rating scales(ALS-FRS) | 6 months
  Changes in ALS-Functional rating scales(ALS-FRS)
Adverse Events(AE) | 6 months
  Incidence & Degree of Adverse Events(AE)

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, M.D., Ph.D, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Cell Therapy Center for Neurologic Disorders, Seoul, Haengdang-dong, Seongdong-gu, South Korea

REFERENCES:
- [Background] Kwon MJ, Baek W, Ki CS, Kim HY, Koh SH, Kim JW, Kim SH. Screening of the SOD1, FUS, TARDBP, ANG, and OPTN mutations in Korean patients with familial and sporadic ALS. Neurobiol Aging. 2012 May;33(5):1017.e17-23. doi: 10.1016/j.neurobiolaging.2011.12.003. Epub 2012 Jan 15. PMID 22244934
- [Background] Koh SH, Baik W, Noh MY, Cho GW, Kim HY, Kim KS, Kim SH. The functional deficiency of bone marrow mesenchymal stromal cells in ALS patients is proportional to disease progression rate. Exp Neurol. 2012 Jan;233(1):472-80. doi: 10.1016/j.expneurol.2011.11.021. Epub 2011 Nov 19. PMID 22119626
- [Background] Koh SH, Huh YM, Noh MY, Kim HY, Kim KS, Lee ES, Ko HJ, Cho GW, Yoo AR, Song HT, Hwang S, Lee K, Haam S, Frank JA, Suh JS, Kim SH. beta-PIX is critical for transplanted mesenchymal stromal cell migration. Stem Cells Dev. 2012 Jul 20;21(11):1989-99. doi: 10.1089/scd.2011.0430. Epub 2012 Jan 26. PMID 22087847
- [Background] Choi MR, Kim HY, Park JY, Lee TY, Baik CS, Chai YG, Jung KH, Park KS, Roh W, Kim KS, Kim SH. Selection of optimal passage of bone marrow-derived mesenchymal stem cells for stem cell therapy in patients with amyotrophic lateral sclerosis. Neurosci Lett. 2010 Mar 19;472(2):94-8. doi: 10.1016/j.neulet.2010.01.054. Epub 2010 Feb 1. PMID 20117176
- [Background] Cho GW, Noh MY, Kim HY, Koh SH, Kim KS, Kim SH. Bone marrow-derived stromal cells from amyotrophic lateral sclerosis patients have diminished stem cell capacity. Stem Cells Dev. 2010 Jul;19(7):1035-42. doi: 10.1089/scd.2009.0453. PMID 20030561
- [Background] Kim H, Kim HY, Choi MR, Hwang S, Nam KH, Kim HC, Han JS, Kim KS, Yoon HS, Kim SH. Dose-dependent efficacy of ALS-human mesenchymal stem cells transplantation into cisterna magna in SOD1-G93A ALS mice. Neurosci Lett. 2010 Jan 14;468(3):190-4. doi: 10.1016/j.neulet.2009.10.074. Epub 2009 Oct 29. PMID 19879334
- [Background] Kwon MS, Noh MY, Oh KW, Cho KA, Kang BY, Kim KS, Kim YS, Kim SH. The immunomodulatory effects of human mesenchymal stem cells on peripheral blood mononuclear cells in ALS patients. J Neurochem. 2014 Oct;131(2):206-18. doi: 10.1111/jnc.12814. Epub 2014 Jul 31. PMID 24995608
- [Background] Oh KW, Moon C, Kim HY, Oh SI, Park J, Lee JH, Chang IY, Kim KS, Kim SH. Phase I trial of repeated intrathecal autologous bone marrow-derived mesenchymal stromal cells in amyotrophic lateral sclerosis. Stem Cells Transl Med. 2015 Jun;4(6):590-7. doi: 10.5966/sctm.2014-0212. Epub 2015 May 1. PMID 25934946
- [Background] Kim HY, Kim H, Oh KW, Oh SI, Koh SH, Baik W, Noh MY, Kim KS, Kim SH. Biological markers of mesenchymal stromal cells as predictors of response to autologous stem cell transplantation in patients with amyotrophic lateral sclerosis: an investigator-initiated trial and in vivo study. Stem Cells. 2014 Oct;32(10):2724-31. doi: 10.1002/stem.1770. PMID 24966156
- See also: collaborator and stem cell provider — http://www.corestem.com
- See also: home page of dementia center in Seoul Seongdong-gu — http://seongdong.seouldementia.or.kr/